CLINICAL TRIAL: NCT04606472
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of SI-B003, a PD-1/CTLA-4 Bispecific Antibody, in Patients With Advanced Solid Tumors
Brief Title: A Study of SI-B003, a PD-1/CTLA-4 Bispecific Antibody, in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI-B003-101
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: Non-small cell lung cancer (NSCLC); Renal cell carcinoma (RCC); Urothelial Cancer (UC); Metastatic colorectal cancer (mCRC); Triple negative breast cancer (TNBC); Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive SI-B003 as intravenous infusion for the first cycle (4 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: SI-B003

INTERVENTIONS:
Drug: SI-B003 — Administration by intravenous infusion.

SUMMARY:
In phase Ia study, the safety and tolerability of SI-B003 in patients with recurrent or metastatic solid tumors will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MAD) for MTD is not reached of SI-B003.

In the phase Ib study, the safety and tolerability of SI-B003 in specific tumors will be further investigated by selecting multiple doses based on the results of phase Ia study or/and the fixed-dose administration method with the closest exposure level, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. The participants could understand and sign the informed consent form, and must participate voluntarily.
2. No gender limit.
3. Age: ≥18 years old and ≤75 years old (phase Ia); ≥18 years old (phase Ib).
4. Expected survival time ≥ 3 months.
5. Histologically or cytologically confirmed recurrent or metastatic solid tumor, clinical stage IIIB/IV, with radiographic or other objective evidence of disease progression after standard therapy; Or subjects were patients with solid tumors that were refractory to treatment, patients with solid tumors that did not have standard treatment, or patients who could not tolerate or had contraindications to standard treatment.
6. For the phase Ib study:

   Cohort_A: Histologically or cytologically confirmed advanced gastric adenocarcinoma (GC) or gastroesophageal junction (GEJ) adenocarcinoma after exposure to platinum-based chemotherapy after receiving only first-line anti-PD-1 (L1) monoclonal antibody during systemic therapy; Cohort_B: Histologically or cytologically confirmed patients with malignant mesothelioma not suitable for surgery;
7. Consent to provide archival tumor tissue or fresh tissue samples of the primary or metastatic tumor, if not available, at the discretion of the investigator (only for stage Ib );
8. At least one measurable lesion that meets the definition of RECIST v1.1 at baseline (only for stage Ib).
9. Patients treated with anti-PD-1 (L1) -containing monoclonal antibody must have progression of resistance after benefit from anti-PD-1 (L1) -containing monoclonal antibody (phase Ib only);
10. Physical fitness score ECOG 0 or 1 point.
11. The adverse reactions of previous antineoplastic therapy returned to CTCAE 5.0 grade ≤1 (except for toxicities without safety risks judged by investigators, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stable with hormone replacement therapy);
12. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
13. The organ function within 7 days prior to the first administration meets the following requirements:

    1. Bone marrow: absolute neutrophil count (ANC) ≥1.5×109/L, hemoglobin ≥90 g/L, platelet count ≥100×109/L (participants with liver cancer ANC ≥75×109/L);
    2. Liver: total bilirubin (TBIL) ≤1.5 ULN (TBIL ≤3 ULN in participants with Gilbert's syndrome, liver cancer or liver metastasis), transaminase (AST/ALT) ≤ 3 ULN (for participants with liver cancer or liver metastasis ≤ 5.0 ULN); for participants with liver cancer or liver metastasis, transaminase ≥ 3 ULN and TBIL ≥ 1.5 ULN must be excluded;
    3. Kidney: Creatinine (Cr) ≤1.5 ULN and creatinine clearance rate (Ccr) ≥ 50mL/min (according to Cockcroft-Gault formula).
14. Female participants with fertility or male participants whose partners are fertile must take effective contraceptive measures from 7 days prior to the first administration to 24 weeks after the administration. Female participants with fertility must have a negative serum/urine pregnancy test in 7 days prior to the first dose.
15. The participants are capable and willing to comply with the visits, treatment plans, laboratory examinations and other study-related procedures stipulated in the study protocol.

Exclusion Criteria:

1. Parenchymal or leptomeningeal metastases with clinical symptoms who were judged by the investigator to be ineligible for enrollment;
2. Participants who participated in any other clinical trial within 28 days before the administration of this trial, except for clinical trials of marketed drugs;
3. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration; oral fluorouracil-like drugs such as S-1, capecitabine, or palliative radiotherapy within 2weeks prior to the first administration.
4. Major surgery (investigator-defined) within 4 weeks before the first dose.
5. In 14 days prior to administration of this study, those who have received systemic corticosteroids (>10mg/day prednisone, or equivalent other corticosteroids) or immunosuppressive therapy should be excluded except for those who have received inhaled or topical corticosteroids, or hormone therapy of physiological replacement dose due to adrenal insufficiency.
6. Pulmonary disease grade ≥3 according to NCI-CTCAE v5.0; Patients with existing interstitial lung disease (ILD).
7. Severe systemic infection occurred within 4 weeks before screening, including but not limited to severe pneumonia caused by fungi, bacteria, viruses, bacteremia, or serious infectious complications.
8. Participants at risk of active autoimmune diseases, or with a history of autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome (polyangiitis granuloma Disease, Graves' disease, rheumatoid arthritis, pituitary inflammation, uveitis), autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barré syndrome), etc. Except for the following conditions: Type I diabetes, hormone replacement therapy for stable hypothyroidism (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo that does not require systemic treatment.
9. Complicated with other malignant tumors within 2 years prior to the first administration, except for cured skin squamous cell carcinoma, basal cell carcinoma, superficial bladder cancer, prostate/cervix/breast carcinoma in situ (only phase Ib).
10. Participants with human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number> 104) or hepatitis C virus (HCV) infection.
11. Participants with poorly controlled hypertension by two kinds of antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg).
12. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, Ⅲ degree atrioventricular block, etc.

    At rest, the QT interval was prolonged (QTc > 450 msec in men or QTc > 470 msec in women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first dose; Patients with New York Heart Association (NYHA) functional class ≥II heart failure.
13. Previous history of allogeneic bone marrow or organ transplantation.
14. Participants who have a history of allergies to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of SI-B003.
15. In the adjuvant (or neoadjuvant) treatment of anthracyclines, the cumulative dose of anthracyclines is> 360 mg/m2.
16. Pregnant or breastfeeding women.
17. Other conditions that the investigator believes that it is not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 28 days after the first dose of SI-B003
  DLTs is assessed according to NCI-CTCAE v5.0 during the first cycle (28 days) and were defined as occurrence of any of the following toxicities if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 28 days after the first dose of SI-B003
  MTD is defined as the dose with the estimated DLT rate closest to the target DLT rate (33%) is selected as the MTD.
  If there are two or more estimated values close to the target DLT rate and the same, when the estimated value is lower than the target DLT rate, choose the higher dose, and when the estimated value is greater than or equal to the target toxicity rate, choose a lower dose.
Phase Ia: Maximum administered dose (MAD) | Up to 28 days after the first dose of SI-B003
  MAD is defined as the maximum administered dose, when MTD is not reached.
Phase Ia: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B003. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B003.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 28 days after the first dose of SI-B003
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B003.

SECONDARY OUTCOMES:
Cmax | Up to 28 days after the first dose of SI-B003
  Maximum serum concentration (Cmax) of SI-B003 will be investigated.
Tmax | Up to 28 days after the first dose of SI-B003
  Time to maximum serum concentration (Tmax) of SI-B003 will be investigated.
T1/2 | Up to 28 days after the first dose of SI-B003
  Half-life (T1/2) of SI-B003 will be investigated.
AUC0-t | Up to 28 days after the first dose of SI-B003
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL | Up to 28 days after the first dose of SI-B003
  Clearance (CL) in the serum of SI-B003 per unit of time will be investigated.
Ctrough | Up to 28 days after the first dose of SI-B003
  Ctrough is defined as the lowest serum concentration of SI-B003 prior to the next dose will be administered.
Adverse Events of special interest (AESI) | Up to approximately 24 months
  AESI is defined as AE that may not be serious but have special meaning or importance for SI-B003.
ADA (Anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of SI-B003 will be evaluated.
NAb (Neutralizing antibody ) | Up to approximately 24 months
  Incidence and titer of NAb of SI-B003 will be evaluated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR was defined as the percentage of participants, who had a CR or PR. The percentage of participants who experienced a confirmed CR or PR is evaluated by investigator and third-party independent medical imaging agency according to RECIST 1.1.
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first. The DOR is evaluated by investigator and third-party independent medical imaging agency according to RECIST 1.1.
Clinical benefit rate (CBR) | Up to approximately 24 months
  CBR was defined as the percentage of participants, who had a CR, PR or SD. The percentage of participants who experienced a confirmed CR, PR or SD is evaluated by investigator and third-party independent medical imaging agency according to RECIST 1.1.
Progression-free survival rate (PFS) | Up to approximately 12 months
  The PFS is defined as the time from the participant's first dose of SI-B003 to the first date of either disease progression or death, whichever occurs first. 6 and 12 months PFS will be evaluated by investigator and third-party independent medical imaging agency according to RECIST 1.1.
Overall survival rate (OS) | Up to approximately 12 months after first dose administration
  12 months OS will be evaluated by investigator and third-party independent medical imaging agency according to RECIST 1.1.
The correlation of PK and clinical efficacy indexes | Up to approximately 24 months
  The correlation of PK parameters (Cmax, AUC0-t, Ctrough, etc.) and clinical efficacy indexes (ORR, CBR, PFS, etc.) will be evaluated.
Evaluation of iORR | Up to approximately 24 months
  iORR will be evaluated by investigator and third-party independent medical imaging agency according to iRECIST 1.1.
Evaluation of iCR | Up to approximately 24 months
  iCR will be evaluated by investigator and third-party independent medical imaging agency according to iRECIST 1.1.
Evaluation of iPR | Up to approximately 24 months
  iPR will be evaluated by investigator and third-party independent medical imaging agency according to iRECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shanghai Central Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan